CLINICAL TRIAL: NCT02320786
Title: Collaborative Power Mobility Innovative Learning OpporTunity (CoPILOT) - A Pilot Study of a New Training Approach (Phase 1)
Acronym: CoPILOT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Networks of Centres of Excellence of Canada (Other); Alzheimer Society of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Promobilia Foundation (Other); Rick Hansen Foundation (Other)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H14-01702
Record Dates: First submitted 2014-12-10; First posted 2014-12-19 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Power Wheelchair; Mild Cognitive Impairment; Spinal Cord Injuries
Keywords: Power mobility; Wheelchair skills training; Spinal Cord Injury
MeSH Terms: conditions — Cognitive Dysfunction; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CoPILOT (Experimental): Experimental group participants will receive structured training in a standard powered wheelchair using the CoPILOT shared control wheelchair technology consisting of 12 hours total training time (one hour, four times per week for three weeks).
  Interventions: Behavioral: CoPILOT
- Standard of Care (No Intervention): Standard of care participants will receive training according to the standard of care in rehabilitation facilities in the Vancouver area in a standard powered wheelchair, consisting of 12 hour protocols in a standard power wheelchair (one hour, four times per week for three weeks).

INTERVENTIONS:
Behavioral: CoPILOT — Participants in both groups will receive twelve hours of training in a standard powered wheelchair however the CoPILOT groups will use remote control technology we have developed. The technology provides the trainer with remote control of wheelchair speed and direction allowing the trainer to override the participant's actions as needed to ensure safe error-free shared controlled wheelchair training. The CoPILOT approach will accommodate varied learning needs, as per adult learning principles, while decreasing trainer input until the participant can complete tasks independently.
  Arms: CoPILOT

SUMMARY:
Losing the ability to walk can lead to fewer opportunities to socialize with friends and family and participate in the community. When this happens, powered wheelchairs can provide access to homes and communities, contributing to health and well-being. Training by a qualified occupational therapist allows an individual to use a powered wheelchair safely and effectively. Learning to drive a powered wheelchair can be difficult, frustrating and time consuming for people with cognitive and physical challenges. In this study, we will ask participants with cognitive impairments to complete training with an occupational therapist using either a shared control wheelchair or training methods according to the standard of care. We believe shared control training, entitled Collaborative Powered mobility Innovative Learning OpporTunity (CoPILOT) will enhance driving skill while maximizing safety learning. CoPILOT has the potential to enable people to participate more in their day to day lives and regain mobility independence.

DETAILED DESCRIPTION:
Background: Powered wheelchairs can improve participation in daily life, increase quality of life, and add 'life to years' for individuals with SCI. Cognitive limitations, associated with advanced age at the time of a spinal cord injury or comorbid traumatic brain injury, impair learning and may prevent an individual from acquiring or maintaining skills necessary to drive a powered mobility device. Standard power wheelchair training, limited by time, equipment and budget constraints, may not meet the learning needs of individuals with cognitive impairment, preventing an individual from obtaining use of a powered wheelchair, impacting independence and quality of life. The total system cost of procuring a power wheelchair can range from $10,000 - $30,000; suboptimal use resulting from inadequate training is a poor use of resources and comes at a substantial social price. The Collaborative Power mobility Innovative Learning OpporTunity (CoPILOT) is a training approach utilizing shared control wheelchair technology and allows a therapist to provide an error-free learning experience for individuals in their own environments, while maintaining safety of the user and the individuals around them. Using shared control technology, the wheelchair user remains in control of the wheelchair while learning to drive, except in cases where the trainer overrides the control (using a remote controlled interface) to maintain safety and provide targeted learning opportunities.

Purpose and Objectives: Our purpose is to obtain pilot data for a larger randomized control trial of a shared control power wheelchair training program (CoPILOT) for improving power wheelchair mobility skills among novice power wheelchair users with comorbid cognitive impairment compared to standard of care. Collection of pilot data is necessary prior to moving forward with a larger randomized controlled trial (RCT).

Hypotheses: We expect the intervention protocol will be feasible for a larger randomized control trial. Compared to the standard of care group, we expect the CoPILOT group will experience significant improvement in power wheelchair skill capacity. We also expect the CoPILOT group will experience improvements in wheelchair skill safety, confidence, capacity for divided attention tasks, and health related quality of life, compared to the standard of care participants.

Methods: Our feasibility study will use an evaluator blind parallel RCT. New power wheelchair users with mild to moderate cognitive impairment will be recruited from the GF Strong or Vancouver General Hospital Spinal Cord Injury patient population. Participants will be randomly assigned to a CoPILOT (shared control training) group or standard of care group. All training will be completed by qualified occupational therapist trainers. Participants in both groups will receive 12 hours of training in a standard powered wheelchair; however, the CoPILOT groups will use remote control technology we have developed. Post-Treatment Qualitative Interviews will be conducted. Questions will be related to protocol administration and use of the CoPILOT approach and shared control technology, including necessary modifications.

ELIGIBILITY:
The following criteria MUST be met in order for the participant to be eligible for the study:

1. Have sustained a spinal cord injury; and
2. Have mild to moderate cognitive impairment (MMSE 18-26); and
3. Be new to powered wheelchairs (no full time driving experience for 3 weeks or more within the past five years) or previously denied a powered wheelchair (due to cognitive impairments impacting ability to learn or inability to learn the required skills); and
4. Be physically able to operate a powered wheelchair joystick.

Participants will not be eligible for the study if ANY of the following criteria are met:

1. Have a visual or hearing impairment which may compromise training safety; OR
2. Do not understand English well enough to complete assessments and/or training.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in Power-mobility Indoor Driving Assessment (PIDA) | Baseline (pre-randomization), 5 weeks (immediate post-intervention)
  The PIDA covers specific tasks required for functional indoor driving, which are specific to the environment (i.e. accessing the bed from the right and left, and approaching the closet and dresser in the bedroom). The PIDA has been evaluated for content and face validity, has good inter-rater (ICC 0.87) and fair intra-rater (ICC 0.67) reliability.55. We aim to explore the potential usefulness of this outcome measure for this population, in this environment, for inclusion in future clinical trials.

SECONDARY OUTCOMES:
Change in Wheelchair Skills Test Questionnaire (WST-P-Q) | Baseline (pre-randomization), 5 weeks (immediate post-intervention)
  The WST-P-Q is a standardized subjective evaluation of the capacity, performance, and confidence for 30 powered wheelchair skills. Total percent scores (0-100%) are calculated for both capacity, performance, and confidence. The WST was selected as a secondary measure because it is a standardized tool for evaluating wheelchair capacity, the primary construct of interest.
Change in Wheelchair-use Confidence Scale (WheelCon-P ) | Baseline (pre-randomization), 5 weeks (immediate post-intervention)
  This measurement for power wheelchair users is a 59-item self-report scale (0-100) with documented reliability and validity. Responses indicate current level of perceived confidence (%) to navigate the physical environment in a wheelchair, perform activities in a wheelchair, problem solve, advocate for specific needs, and manage social situations and emotions. The WheelCon was selected as a secondary outcome measure because confidence for using a wheelchair has been shown to influence wheelchair skills capacity.
Change in Health Utility Index Mark 3 (HUI3) | Baseline (pre-randomization), 5 weeks (immediate post-intervention)
  Health utility measurement is useful in performing cost-utility and cost-effectiveness analyses of new rehabilitation interventions. The HUI3 is a brief questionnaire that asks subjects about their health status, reflected in a single-score measure of health-related quality of life (HRQOL).
Change in The Wheelchair Outcome Measure (WhOM) | Baseline (pre-randomization), 5 weeks (immediate post-intervention)
  The WhOM assess the individual's wheelchair related goals, the importance of those goals, and the satisfaction in their ability to complete those tasks. This will be used to assess goal attainment (performance and satisfaction) following training.
The Wheeling While Talking Test | Baseline (pre-randomization), 5 weeks (immediate post-intervention)
  The Wheeling While Talking Test assesses the individual's ability to complete wheeling tasks under divided attention conditions. This test is being evaluated for use in powered wheelchair studies.
Sensory data | Baseline (pre-randomization), 5 weeks (immediate post-intervention)
  A variety of anonymized sensor data will be collected (not linked to participant files). Data will be used to characterize situations which were deemed unsafe by the trainer, and to analyse steering and intervention behaviours. The following sensor data will be collected from the wheelchair control system (computerized): Joystick movements and button presses (both trainer and participant) and wheelchair movements (odometry). The following sensors data will be collected from sensors attached to the wheelchair: distance to obstacles (laser rangefinders), environmental context (outward looking RGBD cameras), wheelchair movements (accelerometer, gyroscope, compass).

CONTACTS AND LOCATIONS:
Overall Officials: William C Miller, PhD, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Smith EM, Tregobov N, Miller WC. A feasibility study of a shared control powered wheelchair training program for individuals with spinal cord injury. Spinal Cord. 2026 Jan;64(1):40-45. doi: 10.1038/s41393-025-01134-5. Epub 2025 Nov 12. PMID 41225155